CLINICAL TRIAL: NCT01714076
Title: Co-infections in Children Hospitalised for Bronchiolitis: Incidence, Clinical Symptoms and Influence of Cohort Isolation
Brief Title: Co-infections in Children Hospitalised for Bronchiolitis
Status: Completed | Type: Observational
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Principal Investigator, Jolita Bekhof, MD, Princess Amalia Children's Clinic
Other Study IDs: JB-3
Record Dates: First submitted 2012-10-08; First posted 2012-10-25 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum tested for viral agents by PCR-techniques
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort isolation: patients with bronchiolitis are cohorted together irrespective of viral agent diagnosed, thus respiratory syncytial virus (RSV)-positive patient stay in the same room as RSV-negative patients
  Interventions: Other: cohort isolation

INTERVENTIONS:
Other: cohort isolation — all patients hospitalised for bronchiolitis are nursed in one room together, separated from patients without bronchiolitis

SUMMARY:
Observational cohort study in children hospitalized for acute bronchiolitis. Patients are nursed in cohort isolation. Aim is to investigate the incidence and clinical impact of co-infections in this group.

DETAILED DESCRIPTION:
Observational cohort study in children hospitalized for acute bronchiolitis. Patients are nursed in cohort isolation, meaning that all patients admitted for bronchiolitis are cohorted together, irrespective of viral diagnosis. Aim is to investigate the incidence and clinical impact of co-infections in this group.

ELIGIBILITY:
Inclusion Criteria:

* younger than 2 years admitted for bronchiolitis

Exclusion Criteria:

* chronic lung disease congenital heart defect down syndrome

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children < 2 years admitted for bronchiolitis
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
co-infection | approximately 2 weeks
  co-infection acquired during hospitalisation, patient will be followed during hospitalisation and until 1 week after discharge from the hospital, since average duration of hospitalisation in infants with bronchiolitis is 3 days, the time frame will be approximately 2 weeks

SECONDARY OUTCOMES:
clinical severity | approximately 2 weeks
  clinical severity defined as, days of oxygen supplementation, tube feeding, dyspnea score, length of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Jolita Bekhof, MD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands